CLINICAL TRIAL: NCT04660734
Title: Advantages of 3D Printing in the Management of Acetabular Fractures Fixed by the Kocher Langenbeck Approach
Brief Title: Advantages of 3D Printing in the Management of Acetabular Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Mohamed Bouabdellah, MD, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01031972
Record Dates: First submitted 2020-11-11; First posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-11

CONDITIONS: Acetabular Fracture
Keywords: Acetabulum

STUDY DESIGN:
Intervention Model Description: Two techniques for treatment of posterior structure of acetabular fracture
Who Masked: Participant, Outcomes Assessor
Masking Description: Clinical and radiographic results at the last follow-up were evaluated by one surgeon who did not participate in the surgical management of the patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D printing group (Experimental): Group 1 (G1) consisted of 20 patients who underwent preoperative molding of the osteosynthesis plate on a 3D printed model of the pelvis. A preoperative scan of the healthy hemi-pelvis was used to create the 3D-printed model for patients in G1 according to the following three-step methodology: 1) A scanographic acquisition of images was performed using a multi-strip scanner in thin sections. These images were recorded as digital images in the standard medical format of digital imaging and communications ; 2) A digital, 3D model of the pelvis in the stereolithography format was created to digitally treat the 2D images. The individualization of the healthy hemi-pelvis, to which a "mirror effect" was applied allowed for the creation of a symmetrical 3D image, as hemi-pelvises are globally symmetrical. 3) A 3D printer was used to create a physical, 3D-printed model of the affected hemi-pelvis using polylactic acid.
  Interventions: Procedure: Fractures of the posterior structures of the acetabulum treated by fixation using the Kocher-Langenbeck approach.
- conventional technique group (Experimental): Group 2 (G2 or control group) included 23 patients who underwent surgery using the conventional technique.The patients in the control group (G2) underwent surgery following the conventional procedure based on radiographic and CT images with 3D reconstructions.
  Interventions: Procedure: Fractures of the posterior structures of the acetabulum treated by fixation using the Kocher-Langenbeck approach.

INTERVENTIONS:
Procedure: Fractures of the posterior structures of the acetabulum treated by fixation using the Kocher-Langenbeck approach. — Fracture fixation of posterior structures of acetabulum by using the surgical procedure of Kocher-Langenbeck approach

SUMMARY:
Background: Acetabular fractures result from violent trauma, and their incidence has been increasing in recent years. The Kocher-Langenbeck surgical approach is used for the internal fixation of displaced fractures of the posterior structures of the acetabulum. The quality of the reduction and the stability of osteosynthesis directly influence the function of the repaired acetabulum. In the surgical management of acetabulum fractures, 3D printing of a bone model is increasingly used during preoperative planning by trauma surgeons worldwide.

Questions: Is there a difference in the surgical time of the Kocher-langenbeck reduction and fixation of the posterior structures of the acetabulum between 3D printing (which allows for shaping of the reconstruction plate prior to surgery) and the conventional technique? Are there any differences in complications between the two techniques? Are there any short-term differences in the functional and radiographic scores between 3D printing and the conventional technique? Methods: 109 consecutive patients who sustained fractures of the acetabulum were screened for inclusion. 43 patient were studied. The first group (G1) consisted of 20 patients who underwent prior molding of the osteosynthesis plate on a 3D-printed model. The second group (G2 or control group) included 23 patients who underwent surgery using the conventional technique. We compared surgical time, intraoperative blood loss, the difference between pre- and postoperative hemoglobin, and the onset of early infection, paralysis of the sciatic nerve, and deep vein thrombosis.

DETAILED DESCRIPTION:
This randomized, prospective study included 109 consecutive patients who were treated for fractures of the acetabulum between September 2016 and February 2019 at our institution. This study was approved by the ethics committee at our institution and verbal and written informed consent was obtained from all patients. The final analysis included 43 patients (33 males and 10 females) who underwent the Kocher-Langenbeck approach for the reduction and fixation of the posterior structures of the acetabulum.

The patients were divided into two groups. Group 1 (G1) consisted of 20 patients who underwent preoperative molding of the osteosynthesis plate on a 3D printed model of the pelvis. Group 2 (G2 or control group) included 23 patients who underwent surgery using the conventional technique.

All patients were examined in the outpatient department via clinical and radiographic evaluation at 3, 6, 12, and 24 weeks postoperatively, then every 6 months thereafter. A standard radiographic assessment including three views (AP, iliac oblique, and obturator oblique) and a pelvic CT scan were obtained for all patients at the last follow-up visit. The reductions were classified as one of three types: anatomical (residual displacement <1 mm), imperfect (residual displacement 1 to 3 mm), and poor (residual reduction >3 mm). Clinical outcomes were assessed using the modified Harris Hip score. Bone consolidation was obtained in all cases. Clinical and radiographic results at the last follow-up as well as the minimum follow-up duration were evaluated by one surgeon who did not participate in the surgical management of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Fractures of the posterior structures of the acetabulum
* treatment using the Kocher-Langenbeck approach.

Exclusion Criteria:

* age over than 60 years
* treatment approach other than the Kocher-Langenbeck's ( eg orthopedic method)
* open fractures of the pelvis
* fractures of the acetabulum older than 3-weeks
* polytrauma with/or multiple fractures.
* unavailability for follow-up
* insufficient clinical and radiographic data.

Ages: 23 Years to 57 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 109 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Quality of fracture reduction | 30 months with minimum of 18 months
  CT scan displacement of fracture as one of three:
  * Anatomical (residual displacement <1 mm)
  * Imperfect (residual displacement 1 to 3 mm)
  * Poor (residual reduction >3 mm)
radiographic criteria | 30 months with minimum of 18 months
  Matta scoring system a grade of :
  * Excellent :indicates a normal appearance of the hip;
  * Good: mild changes, small osteophytes, moderate (one-millimeter) narrowing of the joint, and minimum sclerosis; a grade of
  * Fair:intermediate changes, moderate osteophytes, moderate (less than 50 per cent) narrowing of the joint, and moderate sclerosis; and a grade of
  * Poor: advanced changes, large osteophytes, severe (more than 50 per cent) narrowing of the joint, collapse or wear of the femoral head, and acetabular wear.
Clinical score | 30 months with minimum of 18 months
  Modified Harris Hip Score includes the pain and function components:
  The maximum score of 91 is multiplied by 1.1 to give a total score out of 100 Modified Hip Harris score
  * Excellent: 90-100
  * Good: 80-90
  * Fair 70-80
  * Poor: <70

CONTACTS AND LOCATIONS:
Overall Officials: Mondher Kooli, PhD, Principal Investigator — Orthopedic and traumatologic department of Charles Nicolle Hospital

IPD SHARING:
Plan to Share IPD: No
No: There is not a plan to make IPD available.

REFERENCES:
- [Background] Wang P, Kandemir U, Zhang B, Fei C, Zhuang Y, Zhang K. The effect of new preoperative preparation method compared to conventional method in complex acetabular fractures: minimum 2-year follow-up. Arch Orthop Trauma Surg. 2021 Feb;141(2):215-222. doi: 10.1007/s00402-020-03472-w. Epub 2020 May 26. PMID 32458075
- [Result] Hsu CL, Chou YC, Li YT, Chen JE, Hung CC, Wu CC, Shen HC, Yeh TT. Pre-operative virtual simulation and three-dimensional printing techniques for the surgical management of acetabular fractures. Int Orthop. 2019 Aug;43(8):1969-1976. doi: 10.1007/s00264-018-4111-8. Epub 2018 Aug 20. PMID 30128670
- [Derived] Bouabdellah M, Bensalah M, Kamoun C, Bellil M, Kooli M, Hadhri K. Advantages of three-dimensional printing in the management of acetabular fracture fixed by the Kocher-Langenbeck approach: randomised controlled trial. Int Orthop. 2022 May;46(5):1155-1163. doi: 10.1007/s00264-022-05319-y. Epub 2022 Feb 1. PMID 35103815